CLINICAL TRIAL: NCT06530550
Title: Exploratory Clinical Study of PI3K Inhibitors in the Treatment of Relapsed/Refractory Indolent T/NK-Cell Lymphomas：An Open, Prospective, Exploratory Clinical Trial
Brief Title: PI3K Inhibitors for the Treatment of Relapsed/Refractory Indolent T/NK-cell Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024026
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, T-Cell; NK-LGL Leukemia; T-LGL Leukemia
Keywords: Indolent T/NK-cell lymphomas; PI3K inhibitor
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PI3K inhibitor (Experimental): Linperlisib 80mg QD orally, or Duvelisib 25mg BID orally
  Interventions: Drug: PI3K inhibitor

INTERVENTIONS:
Drug: PI3K inhibitor — Linperlisib 80mg QD orally, or Duvelisib 25mg BID orally, with a 28-day cycle. Efficacy will be evaluated once per cycle during the first year, and once every two cycles thereafter. Treatment will continue for up to 24 cycles, or until disease progression, lack of response within the first 6 cycles, or the occurrence of intolerable toxicity, whichever occurs first

SUMMARY:
Indolent T/NK-cell lymphomas are a heterogeneous group of lymphoproliferative diseases originating from T/NK cells, characterized by slow growth and proliferation, but currently remain incurable. For indolent T/NK-cell lymphomas that are unresponsive to first-line treatment, there are few treatment options available and the prognosis is poor. This study is an open-label, prospective clinical trial aimed at evaluating the feasibility, efficacy, and safety of PI3K inhibitors in the treatment of relapsed/refractory indolent T/NK-cell lymphomas. Patients will be treated with Linperlisib or Duvelisib, with an expected overall response rate of 60% for PI3K inhibitor treatment.

DETAILED DESCRIPTION:
Plan to enroll 51 patients with relapsed/refractory indolent T/NK-cell lymphomas; they will receive PI3K inhibitor treatment (including Linperlisib 80mg QD orally, or Duvelisib 25mg BID orally, with a 28-day cycle. Efficacy will be evaluated once per cycle during the first year, and once every two cycles thereafter. Treatment will continue for up to 24 cycles, or until disease progression, lack of response within the first 6 cycles, or the occurrence of intolerable toxicity, whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

the proportion of patients whose tumors have not progressed after treatment over a specific period of time. Specifically, DCR includes the percentage of patients who achieve complete response (CR), partial response (PR), and stable disease (SD).

Exclusion Criteria:

Here is the translated text:

1. Subjects who have previously used any PI3K inhibitors;
2. Clinical conditions of dysphagia, malabsorption, or other chronic gastrointestinal diseases that may interfere with compliance and/or absorption of the study drug;
3. Unable to discontinue medications that may prolong the QT interval (such as antiarrhythmic drugs) during the study period;
4. Active viral, bacterial, or fungal infections requiring treatment (e.g., pneumonia);
5. HBV or HCV infection (defined as HBsAg and/or HBcAb positive with HBV DNA copy number ≥ upper limit of normal reference value) or acute or chronic active hepatitis C (HCV) antibody positive;
6. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation, or history of allogeneic bone marrow or hematopoietic stem cell transplantation;
7. Received autologous hematopoietic stem cell transplantation within 90 days before the first dose of study treatment;
8. Presence of severe or uncontrolled cardiovascular disease;
9. Presence of severe concomitant diseases that endanger patient safety or are deemed by the investigator to affect the completion of the study (e.g., uncontrolled hypertension, diabetes, thyroid disease);
10. Pregnant or breastfeeding female patients, or baseline pregnancy test positive for women of childbearing potential;
11. Diagnosed or treated for other malignancies within the past 5 years;
12. Any other condition that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 5 years
  complete remission rate+ partial remission rate

SECONDARY OUTCOMES:
The safety of PI3K inhibitors | up to 5 years
  Incidence of adverse events, serious adverse events and significant adverse event
Complete remession rate | up to 5 years
  Hematological PR was defined as an improvement in blood counts ANC > 0.5 × 109/L; HGB increased by >1 g/dL; PLT > 50 × 109/L
Duration of remission | up to 5 years
  the time from response to progression/death (P/D)
Time to response | up to 5 years
  from the start of treatment to the first observed partial remission
Progression-free survival | up to 5 years
  the time from treatment initiation until disease progression or death
Overall survival | up to 5 years
  The time from the start of treatment to the patient's death from any cause
Disease control rate | up to 5 years
  the proportion of patients whose tumors have not progressed after treatment over a specific period of time. Specifically, DCR includes the percentage of patients who achieve complete response (CR), partial response (PR), and stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No